CLINICAL TRIAL: NCT05464706
Title: Quality of Life After Hepatectomy for Primary Liver Tumors: a Prospective Randomized Clinical Trial on the Role of Supplemental Therapy With Synchrolevels
Brief Title: Study on the Quality of Life (QoL) After Liver Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Humanitas Clinical and Research Center (Other)
Responsible Party: Principal Investigator, Matteo Donadon, Associate Professor of Surgery, Humanitas Clinical and Research Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: QOLILS
Record Dates: First submitted 2022-07-15; First posted 2022-07-19 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Hepatocarcinoma; Cholangiocarcinoma; Quality of Life
MeSH Terms: conditions — Carcinoma, Hepatocellular; Cholangiocarcinoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind: supplement therapy versus placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental)
  Interventions: Dietary Supplement: Synchrolevels
- Control (Placebo Comparator)
  Interventions: Dietary Supplement: Synchrolevels

INTERVENTIONS:
Dietary Supplement: Synchrolevels — Supplement therapy to model the recovery after liver surgery

SUMMARY:
Liver cancer in adult men is the fifth most frequently diagnosed cancer worldwide, and is the second leading cause of cancer-related death in the world. To date, liver surgery is the treatment of choice for those patients with resectable disease. However, still today the proportion of resectable patients is limited due to a large proportion of patients presenting with advances disease. For these patients, the treatment consists of systemic chemotherapy, which unfortunately is associated with median survival of 12 months. The choice of the appropriate treatment scheme adheres to the standard guidelines based on the results of clinical trials. Of note, in case of HCC and MFCCC very few international approved therapeutic guidelines are available. In particular, there is no agreement among specialists about the use of chemotherapy as adjuvant treatment after hepatic resection for HCC or MFCCC. An important aspect of the postoperative "adjuvant therapy" is the possibility to enhance the recovery after the operation. Indeed, the possibility to accelerate the functional recovery in a patient who receives a major cancer operation is of paramount importance. In this sense, having a product that might help the patients' recovery should be one of the priorities of the medical and pharmaceutical industry. To our knowledge, there are no previous studies that investigated such an important aspect.

DETAILED DESCRIPTION:
Liver cancer in adult men is the fifth most frequently diagnosed cancer worldwide, and is the second leading cause of cancer-related death in the world. In adult women, it is the seventh most commonly diagnosed cancer and the sixth leading cause of cancer death. The two main types of liver cancer are hepatocellular carcinoma (HCC) and mass-forming cholangiocarcinoma (MFCCC). The annual overall incidence is approximately 70 and 2 per 100,000 inhabitants for HCC and MFCCC respectively.

To date, liver surgery is the treatment of choice for those patients with resectable disease. For some other patients, with specific tumor features, liver transplantation may be applied with good results. However, still today the proportion of resectable or transplantable patients is limited due to a large proportion of patients presenting with advances disease. For these patients, the treatment consists of systemic chemotherapy, which unfortunately is associated with median survival of 12 months. The choice of the appropriate treatment scheme adheres to the standard guidelines based on the results of clinical trials. Of note, in case of HCC and MFCCC very few international approved therapeutic guidelines are available. In particular, there is no agreement among specialists about the use of chemotherapy as adjuvant treatment after hepatic resection for HCC or MFCCC. In other words, in the actual clinical practice a patient operated for HCC or MFCCC generally does not receive postoperative adjuvant chemotherapy.

Another important aspect of the postoperative adjuvant therapy is the possibility to enhance the recovery after the operation. Indeed, the possibility to accelerate the functional recovery in a patient who receives a major cancer operation is of paramount importance. In this sense, having a product that might help the patients' recovery should be one of the priorities of the medical and pharmaceutical industry. To our knowledge, there are no previous studies that investigated such an important aspect.

Synchro Levels consists of a supplemental nutritional therapy that has been present on the market for more than 15 years. Some studies reported its safety and efficacy in patients with different advanced solid tumors showing an unexpected rate of partial response. However, very few data are available on its role in improving the patients' performance status and the quality of life. This research project aims to test the role of Synchro Levels in enhancing the functional recovery of patients submitted to hepatectomy for HCC or MFCCC.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age ≥ 18 years old
* First diagnosis and first hepatectomy for HCC or MFCCC

Exclusion Criteria:

* Refute to sign the informed consent
* Age < 18 years old
* Indication to perform adjuvant (postoperative) chemotherapy
* Any psychological or psychiatric condition that might compromise the patients' compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Quality of life after liver surgery | 6 months
  Quality of life (recovery after liver surgery) measured by using the European form SF36. The 36-Item Short Form Survey (SF-36) is an oft-used, well-researched, self-reported measure of health. It comprises 36 questions which cover eight domains of health.

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Research Hospital, Rozzano, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No